CLINICAL TRIAL: NCT01182753
Title: Randomised Trial of Proton vs. Carbon Ion Radiation Therapy in Patients With Low and Inter-mediate Grade Chondrosarcoma of the Skull Base, Clinical Phase III Study
Brief Title: Trial of Proton Versus Carbon Ion Radiation Therapy in Patients With Low and Inter-mediate Grade Chondrosarcoma of the Skull Base
Acronym: CSP12C
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Dr. Dr. J. Debus, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS.P.12C
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Chondrosarcoma
Keywords: Chondrosarcoma; Radiation; carbon ion
MeSH Terms: conditions — Chondrosarcoma | interventions — Heavy Ion Radiotherapy; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm A (carbon ion therapy):
  Total dose to the PTV2 - 45 Gy E in 3 Gy E /d, 4 - 6 days a week, 15 fractions Total dose to the PTV1 - 60 Gy E ± 5%, further 4 - 6 fractions a 3 Gy E.
  Interventions: Radiation: carbon ion therapy
- B (Active Comparator): Arm B (proton therapy):
  Total dose to the PTV2 - 50 to 56 Gy E in 2 Gy E /d, 4 - 6 days a week, 25 - 28 fractions Total dose to the PTV1 - 70 Gy E ± 5%, further 6 - 10 fractions a 2 Gy E.
  Interventions: Radiation: proton therapy

INTERVENTIONS:
Radiation: carbon ion therapy — Arm A (carbon ion therapy):
  Total dose to the PTV2 - 45 Gy E in 3 Gy E /d, 4 - 6 days a week, 15 fractions Total dose to the PTV1 - 60 Gy E ± 5%, further 4 - 6 fractions a 3 Gy E.
  Arms: A
Radiation: proton therapy — Arm B (proton therapy):
  Total dose to the PTV2 - 50 to 56 Gy E in 2 Gy E /d, 4 - 6 days a week, 25 - 28 fractions Total dose to the PTV1 - 70 Gy E ± 5%, further 6 - 10 fractions a 2 Gy E.
  Arms: B

SUMMARY:
The study is a prospective randomised clinical phase III trial. Proton therapy is the gold standard in the treatment of low and intermediate grad chondrosarcomas of the skull base. However, high-LET beams such as carbon ions theoretically offer biologic advantages by enhanced biologic effectiveness in slow-growing tumors. Up until now it was impossible to compare two different particle therapies, i.e. proton and carbon ion therapy directly with each other. The aim of this study is to find out, whether the biological advantages of carbon ion therapy mentioned above can also be clinically confirmed.

DETAILED DESCRIPTION:
The study is a prospective randomised clinical phase III trial. The trial will be carried out at Heidelberger Ionenstrahl-Therapie (HIT) centre as monocentric trial.

Proton therapy is the gold standard in the treatment of low and intermediate grad chondrosarcomas of the skull base. However, high-LET beams such as carbon ions theoretically offer biologic advantages by enhanced biologic effectiveness in slow-growing tumors. Up until now it was impossible to compare two different particle therapies, i.e. proton and carbon ion therapy directly with each other. The aim of this study is to find out, whether the biological advantages of carbon ion therapy mentioned above can also be clinically confirmed.

Patients with skull base chondrosarcomas will be randomised to either proton or carbon ion radiation therapy. As a standard, patients will undergo non-invasive, rigid immobilization and target volume definition will be carried out based on CT and MRI data. The biologically isoeffective target dose to the PTV in carbon ion treatment will be 60 Gy E ± 5% and 70 Gy E ± 5% (standard dose) in proton therapy respectively. The 5 year local-progression free survival (LPFS) rate will be analysed as primary end point. Overall survival, progression free and metastasis free survival, patterns of recurrence, local control rate and morbidity are the secondary end points. Plan quality is also a matter of interest.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Score ≥60%
* Age >18 years and <80 years
* Informed consent signed by the patient
* Histological confirmation of low/ intermediate grade chondrosarcoma with infiltration of the skull base.

Exclusion Criteria:

* Inability to understand the aims of the study, no informed consent
* Prior RT of skull base region
* Other malignancies with disease-free interval < 5 years (excepting pre-cancerous lesions)
* Participation in another trial
* Pregnancy
* Simultaneous CHT or Immunotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2010-08; Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Local-Progression Free Survival (LPFS) | 5 years
  The primary objective of this study is to evaluate, if the innovative carbon ion therapy in chondrosarcomas is not relevantly inferior to the standard proton treatment with respect to the 5 year LPFS rate defined as time from the randomisation to observed local reccurrence. It is assumed that the LPFS rate for the proton therapy is 90%.

SECONDARY OUTCOMES:
Survival | 12 years
  Assessment of overall survival, progression free and metastasis free survival.
Toxicity | 12 years
  Acute and late toxicity will be analysed according to Common Terminology Criteria for Adverse Events: CTCAE V4.0 for acute side effects and RTOG/EORTC for late reaction.
Patterns of recurrence and local control rate | 5 years
  Local recurrences will be confirmed radiologically and histologically whenever possi-ble. At least two medical doctors (radiation oncologist and/or radiologist) will be re-quired to judge of the recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD PhD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Im Neuenheimer Feld 400, Germany

REFERENCES:
- [Background] Schulz-Ertner D, Nikoghosyan A, Hof H, Didinger B, Combs SE, Jakel O, Karger CP, Edler L, Debus J. Carbon ion radiotherapy of skull base chondrosarcomas. Int J Radiat Oncol Biol Phys. 2007 Jan 1;67(1):171-7. doi: 10.1016/j.ijrobp.2006.08.027. Epub 2006 Oct 23. PMID 17056193
- [Background] Munzenrider JE, Liebsch NJ. Proton therapy for tumors of the skull base. Strahlenther Onkol. 1999 Jun;175 Suppl 2:57-63. doi: 10.1007/BF03038890. PMID 10394399
- [Background] Ares C, Hug EB, Lomax AJ, Bolsi A, Timmermann B, Rutz HP, Schuller JC, Pedroni E, Goitein G. Effectiveness and safety of spot scanning proton radiation therapy for chordomas and chondrosarcomas of the skull base: first long-term report. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1111-8. doi: 10.1016/j.ijrobp.2008.12.055. Epub 2009 Apr 20. PMID 19386442
- [Background] Hug EB, Slater JD. Proton radiation therapy for chordomas and chondrosarcomas of the skull base. Neurosurg Clin N Am. 2000 Oct;11(4):627-38. PMID 11082173
- [Background] Hug EB, Loredo LN, Slater JD, DeVries A, Grove RI, Schaefer RA, Rosenberg AE, Slater JM. Proton radiation therapy for chordomas and chondrosarcomas of the skull base. J Neurosurg. 1999 Sep;91(3):432-9. doi: 10.3171/jns.1999.91.3.0432. PMID 10470818
- [Background] Weber DC, Rutz HP, Pedroni ES, Bolsi A, Timmermann B, Verwey J, Lomax AJ, Goitein G. Results of spot-scanning proton radiation therapy for chordoma and chondrosarcoma of the skull base: the Paul Scherrer Institut experience. Int J Radiat Oncol Biol Phys. 2005 Oct 1;63(2):401-9. doi: 10.1016/j.ijrobp.2005.02.023. PMID 16168833
- [Derived] Nikoghosyan AV, Rauch G, Munter MW, Jensen AD, Combs SE, Kieser M, Debus J. Randomised trial of proton vs. carbon ion radiation therapy in patients with low and intermediate grade chondrosarcoma of the skull base, clinical phase III study. BMC Cancer. 2010 Nov 5;10:606. doi: 10.1186/1471-2407-10-606. PMID 21050498